CLINICAL TRIAL: NCT01810159
Title: Integrated Collaborative Care for Substance Use Disorders
Acronym: SUMMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01DA034266 (NIH)
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Substance Use Disorders
Keywords: substance use disorders; implementation science; collaborative care; opiate disorders; alcohol disorders
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders | interventions — Educational Status; Health Resources

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: We used an R software random number generator to randomly assign eligible participants to either CC or usual care. We used a concealed randomization protocol where neither participant nor researcher (outside of the statistician doing the randomization) was aware of the randomization until after the baseline interview. None of the participants or providers was blinded to treatment allocation after randomization. Interviewers were blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICC (Experimental): Integrated collaborative care
  Interventions: Other: Integrated collaborative care
- E&R (Active Comparator): Education and Resources--enhanced usual care
  Interventions: Other: Education and Resources

INTERVENTIONS:
Other: Integrated collaborative care
  Arms: ICC
Other: Education and Resources
  Arms: E&R

SUMMARY:
Primary care settings (PCS) are a missed opportunity for delivering evidence-based treatments for opiate and alcohol-use disorders (OAUD). The investigators propose to evaluate the costs and effectiveness of two strategies to increase the delivery of OAUD treatments in PCS, integrated collaborative care (ICC) and education and resources (E&R). The investigators hypothesize that ICC will be more effective than E&R in promoting A. Implementation outcomes B. Service system outcomes and C. Patient outcomes.

Results from our study will help providers choose between two different strategies and advance the field of implementation research.

DETAILED DESCRIPTION:
Most individuals with opiate and alcohol-use disorders (OAUD) do not receive treatment. Primary care is an ideal setting in which to deliver OAUD treatment, yet evidence-based OAUD treatment is rarely provided.

Barriers to delivery include insufficient organizational support and lack of provider role models and clinical support. The investigators propose to evaluate the effectiveness of two strategies for increasing use of evidence-based treatment for OAUD within primary care: integrated collaborative care (ICC) and education and resources (E&R). While both strategies provide primary care practices with the same clinical information, ICC addresses these barriers by including organizational and technical support for delivering evidence-based care. ICC is grounded in the chronic care model and includes a behavioral health provider working as part of the care team.

Essential elements of ICC strategy include a decision support component to help providers with complex patients, and a restructuring of the delivery and clinical information systems to support the delivery of evidence-based care. Our approach to implementing ICC is based on the organizational transformation model and quality improvement. The investigators define the E&R strategy as providing printed educational materials and access to resources along with provider education. Both strategies are designed to increase the delivery of two evidence-based practices: motivational enhancement therapy and medication assisted therapy.

The investigators propose a 5-year mixed methods study and will conduct a RCT, with randomization occurring at the level of the care team and patient. The investigators partner with 5 Venice Family Clinic (VFC) clinics, two hospitals in LA County, and COPE Health Solutions. VFC is a large federally qualified health center (FQHC) and the largest free clinic in the United States. Our approach includes document review, focus groups, interviews, and surveys for obtaining data on the adoption process and implementation outcomes; analysis of patient records and patient surveys on service system and patient outcomes; and analysis of provider financial records and patient records and surveys for estimating costs. The investigators will enroll 400 patients with an OAUD diagnosis and follow them at 3 and 12 months. Our specific aims are: 1) To measure the process and extent of ICC and E&R implementation; 2) To test the effectiveness of ICC compared to an E&R strategy in promoting A. Implementation outcomes B. Service system outcomes and C. Patient outcomes; and 3) To estimate provider costs for each strategy. The investigators define implementation outcomes as measures of the acceptability, adoption, appropriateness, feasibility, and sustainability of evidence-based OAUD treatment. The investigators define service system outcomes as 1) process measures of treatment quality and 2) treatment co-morbidities. The investigators define patient outcomes as hospital readmissions, OAUD outcomes, patient functioning, negative consequences from substance use, and unmet need. The investigators define cost outcomes as start-up costs, operating costs and medical/psychiatric cost offsets.

ELIGIBILITY:
Inclusion Criteria:

* opiate or alcohol use disorder
* not currently in substance use disorder treatment
* past 30 day use of alcohol or opioids
* English or Spanish speaking

Exclusion Criteria:

* co-morbid severe mental illness
* medically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2014-06; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
unmet need | past 6 months
  Of those identified as screening positive for an opiate or alcohol use disorder, proportion who did not receive treatment for their substance use
abstinent from alcohol and opioid use, past 30 days | past 30 days
  change in abstinence from alcohol and opioid use between baseline and 6 month follow up
negative consequences related to substance use | past 3 months
  SIP-AD frequency questionnaire
Functioning | past 4 weeks
  change in SF-12 between baseline and follow up
Engagement | 30 days of initiation
  Proportion with at least 2 SUD-related visits within 30 days of initiation, Washington Circle
initiation | Within 14 days of index visit
  Washington Circle initiation indicator--at least one SUD-related visit within 14 days of index visit
heavy alcohol use | 6 months
  among people at baseline with heavy alcohol use, proportion with heavy alcohol use in past 30 days

SECONDARY OUTCOMES:
Proportion initiating Brief therapy | 6 months
  Proportion initiating brief therapy within 6 months
Proportion initiating MAT | 6 months
  Proportion initiating MAT within 6 months, among those eligible for MAT, and if N's are large enough, stratified by type of MAT
abstinence from alcohol, opioids and all other drugs in the previous 30 days | collected at six months at the past 30 days
  abstinence from alcohol, opioids and all other drugs in the past 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Venice Family Clinic-Simms Mann Health Center, Santa Monica, California
  - Venice Family Clinic-Rose lAvenue, Venice, California

REFERENCES:
- [Derived] Hunter SB, Ober AJ, McCullough CM, Storholm ED, Iyiewuare PO, Pham C, Watkins KE. Sustaining alcohol and opioid use disorder treatment in primary care: a mixed methods study. Implement Sci. 2018 Jun 18;13(1):83. doi: 10.1186/s13012-018-0777-y. PMID 29914524
- [Derived] Watkins KE, Ober AJ, Lamp K, Lind M, Setodji C, Osilla KC, Hunter SB, McCullough CM, Becker K, Iyiewuare PO, Diamant A, Heinzerling K, Pincus HA. Collaborative Care for Opioid and Alcohol Use Disorders in Primary Care: The SUMMIT Randomized Clinical Trial. JAMA Intern Med. 2017 Oct 1;177(10):1480-1488. doi: 10.1001/jamainternmed.2017.3947. PMID 28846769
- [Derived] Ober AJ, Watkins KE, Hunter SB, Lamp K, Lind M, Setodji CM. An organizational readiness intervention and randomized controlled trial to test strategies for implementing substance use disorder treatment into primary care: SUMMIT study protocol. Implement Sci. 2015 May 8;10:66. doi: 10.1186/s13012-015-0256-7. PMID 25951953